CLINICAL TRIAL: NCT06561243
Title: Ibrutinib and Acalabrutinib Use and Risk of Atrial Fibrillation in Patients With Chronic B-cell Malignancies
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Joachim ALEXANDRE, Professor, University Hospital, Caen
Other Study IDs: Pharmaco072424
Record Dates: First submitted 2024-07-24; First posted 2024-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Chronic B-cell Malignancies; BTK Inhibitors; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — ibrutinib; acalabrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ibrutinib: Adult patients with a chronic B-cell malignancy exposed to ibrutinib
  Interventions: Drug: BTK inhibitor (Ibrutinib or Acalabrutinib)
- Acalabrutinib: Adult patients with a chronic B-cell malignancy exposed to acalabrutinib
  Interventions: Drug: BTK inhibitor (Ibrutinib or Acalabrutinib)

INTERVENTIONS:
Drug: BTK inhibitor (Ibrutinib or Acalabrutinib) — Adult patients with a chronic B-cell malignancy included in this study will be separate into 2 groups according to the BTK inhibitor (ibrutinib and acalabrutinib)

SUMMARY:
Background. Ibrutinib and acalabrutinib are both associated with an increased risk of atrial fibrillation (AF) but AF comparative risk between these 2 BTK inhibitors (BTKis) remains largely unknown.

Objectives. Our aim was to examine the risk of developing incident AF with ibrutinib exposure compared with acalabrutinib exposure.

Methods. Using the TriNetX research network database, authors will conduct a retrospective cohort analysis of deidentified, aggregate adult patients with chronic B-cell malignancies and exposed to ibrutinib or acalabrutinib. Patients will be divided into 2 groups based on ibrutinib or acalabrutinib exposure. After propensity score matching (PSM), hazard ratios (HRs) and their associated 95% confidence intervals (CIs) will be used to compare AF risk during follow-up between the matched 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* diagnose with chronic B-cell malignancies using ICD-10-CM codes C91 (lymphoid leukemia), C88.0 (Waldenström macroglobulinemia), C83.1 (mantle cell lymphoma), C81-C96 (malignant neoplasms of lymphoid, hematopoietic and related tissue) or C95 (leukemia of unspecified cell type)
* expose to ibrutinib or acalabrutinib determined by the Anatomical Therapeutic Chemical codes

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients - diagnose with chronic B-cell malignancies expose to ibrutinib or acalabrutinib in the TrinetX database
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Risk of incident atrial fibrillation in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort. | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code I48 will be used to identify AF during follow-up

SECONDARY OUTCOMES:
Risk of incident atrial fibrillation in patients exposed to ibrutinib compared with those exposed to acalabrutinib in a matched cohort restricted to patients aged ≤75 and to patients aged >75 | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code I48 will be used to identify AF during follow-up
Risk of incident atrial fibrillation in patients exposed to ibrutinib compared with those exposed to acalabrutinib in a matched cohort categorized according their baseline cardiovascular risk level for developing AF | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code ill be used to identify AF during follow-up
Risk of all-cause mortality in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort | from the introduction of the BTK inhibitor and up to 120 months
  death from any cause during follow-up
Risk of incident intra-cerebral hemorrhage in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code ill be used to identify intra-cerebral hemorrhage during follow-up
Risk of incident major bleeding in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code ill be used to identify major bleeding during follow-up
Risk of incident hypertension in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code ill be used to identify hypertension during follow-up
Risk of incident MACE (composite) in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code ill be used to identify MACE (composite of acute myocardial infraction, ischemic stroke or thromboembolism and heart failure) during follow-up
Risk of incident ventricular tachycardia/ventricular fibrillation/cardiac arrest (composite) in patients exposed to ibrutinib compared with those exposed to acalabrutinib in the whole matched cohort | from the introduction of the BTK inhibitor and up to 120 months
  ICD-10-CM code ill be used to identify VT/VF/cardiac arrest (composite of ventricular tachycardia, ventricular fibrillation and cardiac arrest) during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Department of Pharmacology, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No
Actually, data from TrinetX are only freely available for health care organizations participating to the health research network database.

REFERENCES:
- [Derived] Alexandre J, Font J, Lenormand T, Chantepie S, Bardet H, Damaj G, Dolladille C, Legallois D, Da-Silva A, Milliez P, Bisson A, Fauchier L. Ibrutinib and acalabrutinib use and risk of incident atrial fibrillation: a propensity-matched analysis. Exp Hematol Oncol. 2025 Mar 4;14(1):29. doi: 10.1186/s40164-025-00619-6. PMID 40038806